CLINICAL TRIAL: NCT01810809
Title: Hip Viscosupplementation: What is the Best Dosage?
Acronym: Hip VS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0255/10
Record Dates: First submitted 2013-03-11; First posted 2013-03-14 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Hip; Viscosupplementation; Clinical Trial
MeSH Terms: conditions — Osteoarthritis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Articular Lavage (Active Comparator): Patients from Group Zero will receive articular lavage with saline injection
  Interventions: Procedure: articular lavage with saline injection
- Group 1 (Experimental): Patients from Group 1 will receive articular lavage with saline injection and viscosupplementation with 2ml (1 ampoule) of Hylan GF-20
  Interventions: Procedure: articular lavage with saline injection; Drug: 1 ampoule of Hylan GF-20
- Group 2 (Experimental): Patients from Group 2 will receive articular lavage with saline injection and viscosupplementation with 4ml (2 ampoules) of Hylan GF-20
  Interventions: Procedure: articular lavage with saline injection; Drug: 2 ampoules of Hylan GF-20
- Group 3 (Experimental): Patients from Group 3 will receive articular lavage with saline injection and viscosupplementation with 6ml (3 ampoules) of Hylan GF-20
  Interventions: Procedure: articular lavage with saline injection; Drug: 3 ampoules of Hylan GF-20

INTERVENTIONS:
Procedure: articular lavage with saline injection — Patients will receive articular lavage with saline injection
Drug: 1 ampoule of Hylan GF-20 — Patients will receive viscosupplementation with 2ml (1 ampoule) of Hylan GF-20
  Other Names: 1 ampole of Synvisc Classic
  Arms: Group 1
Drug: 2 ampoules of Hylan GF-20 — Patients will receive viscosupplementation with 4ml (2 ampoules) of Hylan GF-20
  Other Names: 2 ampoles of Synvisc Classic
  Arms: Group 2
Drug: 3 ampoules of Hylan GF-20 — Patients will receive viscosupplementation with 6ml (3 ampoules) of Hylan GF-20
  Other Names: 3 ampoules of Synvisc Classic
  Arms: Group 3

SUMMARY:
Intraarticular injections have long been used to treat osteoarthritis. Viscosupplementation is a relatively new approach comprising the injection of hyaluronic acid into diarthrodial joints. The dosis regimen is well established for the knee joint, but there is still no consensus regarding the optimal dosage for hip viscosupplementation. Our objective is to determine the optimal dosis for hip viscosupplementation

DETAILED DESCRIPTION:
Intraarticular injections have long been used to treat osteoarthritis. Viscosupplementation is a relatively new approach comprising the injection of hyaluronic acid into diarthrodial joints. Any osteoarthritic joint is eligible to this treatment modality, but the great majority of studies are for knee viscosupplementation. The dosis regimen is well established for the knee joint, but there is still no consensus regarding the optimal dosage for hip viscosupplementation. We will prospectively enroll 80 patients with hip osteoarthritis and will randomize them into four groups: Group zero will receive joint lavage with saline injection. Group 1 will receive joint lavage with saline injection and 2 ml of Hylan GF-20 (1 ampoule of Synvisc Classic®). Group 2 will receive joint lavage with saline injection and 4 ml of Hylan GF-20 (2 ampoules of Synvisc Classic®). Group 3 will receive joint lavage with saline injection and 6 ml of Hylan GF-20 (3 ampoules of Synvisc Classic®). The Visual Analogic Scale of Pain (VAS), the Western Ontario and McMaster Universities Index (WOMAC®), and Lequesne questionnaires were completed at baseline and at Weeks 1, 4, 12, and 24. Our objective is to determine the optimal dosis for hip viscosupplementation

ELIGIBILITY:
Inclusion Criteria:

* Met the American College of Rheumatology criteria for hip osteoarthritis
* No hip intraarticular injections in the last 6 months

Exclusion Criteria:

- Severe reaction to the procedure

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-06 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
WOMAC | 6 months
  Pain and function assessment with WOMAC questionaire
VAS | 6 months
  Pain assessment with Visual Analogic Scale (VAS)
Lequesne | 6 months
  Pain and function assessment with Lequesne questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo C de Campos, MD, Principal Investigator — FMUSP
Locations (1):
- Instituto de Ortopedia e Traumatologia HC-FMUSP, São Paulo, São Paulo, Brazil